CLINICAL TRIAL: NCT00231868
Title: A Pilot Phase II Trial of Radiation Therapy "Sandwiched" Between Paclitaxel and Carboplatin in Patients With Uterine Papillary Serous Carcinoma
Brief Title: A Study of Radiation Therapy and Paclitaxel and Carboplatin in Patients With Uterine Papillary Serous Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Yi-Shin Kuo, Attending, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-09-227
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Uterine Cancer
Keywords: Uterine Papillary Serous Carcinoma; UPSC; Radiation Therapy; Chemotherapy
MeSH Terms: conditions — Uterine Neoplasms | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Drug:Carboplatin and Paclitaxel and Radiation: Pelvic Radiation Therapy
  Interventions: Drug: Carboplatin and Paclitaxel and Pelvic Radiation Therapy; Procedure: Carboplatin and Paclitaxel and Pelvic Radiation Therapy; Drug: Carboplatin and Paclitaxel and Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin and Paclitaxel and Pelvic Radiation Therapy — Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
Procedure: Carboplatin and Paclitaxel and Pelvic Radiation Therapy — Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
Drug: Carboplatin and Paclitaxel and Radiation Therapy — Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles

SUMMARY:
Combination chemo/radiotherapy trials in advanced/recurrent endometrial cancer are ongoing. The optimal radiation modality, chemotherapeutic agents, and sequence of these regimens for the treatment of UPSC are yet to be established. A retrospective review of 16 patients treated at our institution with the sequential use of radiation "sandwiched" between paclitaxel/platinum chemotherapy found only one patient to have recurred at 16 months with a median follow-up of 15 months (range 6-33 months). The regimen was well tolerated. Eight of the sixteen patients (50%) developed grade 3 neutropenia following cycle 4 of chemotherapy, two of which required a 1 week treatment delay. There were no cases of grade 3 or 4 thrombocytopenia noted. There was no febrile neutropenia and no hospital admissions for toxicity. There were no observed grade 3 or 4 non-hematologic toxicities. With the median follow up of 15 months, we have not observed late toxicities.

Given these favorable preliminary findings, supported by recently published data documenting efficacy of the "sandwich" multimodality technique in other difficult uterine malignancies (malignant mixed mullerian tumors), we propose to study this combination of chemotherapy and radiation prospectively. Our aim is to better evaluate patterns of recurrence and possible benefits in progression-free and overall survival.

DETAILED DESCRIPTION:
Uterine papillary serous carcinoma (UPSC) is an uncommon, but aggressive variant of endometrial carcinoma that has a high recurrence rate and poor response to therapy. It has a propensity to metastasize throughout the abdomen, similar to serous carcinoma of the ovary. In fact, many patients with disease apparently confined to the uterus have microscopic intra-abdominal spread at the time of diagnosis. Recurrences are common both in the pelvis as well as in the upper abdomen.

After staging and debulking of gross disease, adjuvant radiation therapy is recommended to treat patients with endometrial carcinoma at high risk for recurrent disease. High-risk features include histologic cell type, grade, depth of myometrial invasion, cervical extension, lymph-vascular invasion, adnexal involvement, intraperitoneal spread, positive peritoneal cytology, and positive lymph nodes. Pelvic radiation can limit local recurrences to less than 6.5%. However, approximately 25-30% of patients with high-risk features who receive radiation recur with distant metastases. Even patients treated with whole abdominal irradiation are at risk for extra-abdominal recurrences with progression-free intervals of 7 to 8 months.

Adjuvant chemotherapeutic regimens have been studied in high-risk endometrial cancers, but none have demonstrated a survival advantage. Doxorubicin, in combination with platinum, has a reported 42% response rate, but a high toxicity profile. Paclitaxel has an overall response rate of 36% in patients with advanced and recurrent endometrial cancer. Platinum-based chemotherapies have a 28-42% response rate.

Retrospective studies in patients with UPSC have demonstrated response rates of up to 35% in patients with multiagent chemotherapy. In one study, a median progression-free interval of 30 months was observed in patients treated with paclitaxel and platinum in the adjuvant and recurrent settings. Based on these findings and the similarities and clinical success of paclitaxel/platinum therapy in patients with ovarian serous carcinoma, this combination warrants further investigation in a prospective manner in patients with UPSC.

Combination chemo/radiotherapy trials in advanced/recurrent endometrial cancer are ongoing. The optimal radiation modality, chemotherapeutic agents, and sequence of these regimens for the treatment of UPSC are yet to be established. A retrospective review of 16 patients treated at our institution with the sequential use of radiation "sandwiched" between paclitaxel/platinum chemotherapy found only one patient to have recurred at 16 months with a median follow-up of 15 months (range 6-33 months). The regimen was well tolerated. Eight of the sixteen patients (50%) developed grade 3 neutropenia following cycle 4 of chemotherapy, two of which required a 1 week treatment delay. There were no cases of grade 3 or 4 thrombocytopenia noted. There was no febrile neutropenia and no hospital admissions for toxicity. There were no observed grade 3 or 4 non-hematologic toxicities. With the median follow up of 15 months, we have not observed late toxicities.

Given these favorable preliminary findings, supported by recently published data documenting efficacy of the "sandwich" multimodality technique in other difficult uterine malignancies (malignant mixed mullerian tumors), we propose to study this combination of chemotherapy and radiation prospectively. Our aim is to better evaluate patterns of recurrence and possible benefits in progression-free and overall survival.

Surrogate endpoint biomarkers such as ER/PR, HER2/Neu and p53 will be correlated with prognosis. In addition, fresh frozen tissue will be banked for future cDNA microarray analyses of UPSC tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented uterine papillary serous carcinoma (UPSC) with no visible residual disease.
2. Surgical staging to include total abdominal hysterectomy, bilateral salpingo-oophorectomy, peritoneal washings, and lymph node samplings.
3. Age > 18 years.
4. ECOG performance status of < 2.
5. Written voluntary informed consent.

Exclusion Criteria:

1. Patient has impairment of hepatic, renal or hematologic function as defined by the following baseline laboratory values:

   1. Serum SGOT and /or SGPT > 2.5 times the institutional upper limit of normal
   2. Total serum bilirubin > 1.5 mg/dl
   3. History of chronic or active hepatitis
   4. Serum creatinine > 2.0 mg/dl
   5. Platelets < 100,000/mm3
   6. Absolute neutrophil count (ANC) < 1500/mm3
   7. Hemoglobin < 8.0 g/dl (the patient may be transfused prior to study entry)
2. Patient has severe or uncontrolled concurrent medical disease (eg. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
3. Patient has been treated with myelosuppressive chemotherapy within three weeks prior to study entry.
4. Patient with any prior chemotherapy or radiotherapy for pelvic malignancy.
5. Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at the time of study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2001-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Einstein, M.D., M.S., Principal Investigator — Montefiore Medical Center and Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Einstein MH, Frimer M, Kuo DY, Reimers LL, Mehta K, Mutyala S, Huang GS, Hou JY, Goldberg GL. Phase II trial of adjuvant pelvic radiation "sandwiched" between combination paclitaxel and carboplatin in women with uterine papillary serous carcinoma. Gynecol Oncol. 2012 Jan;124(1):21-5. doi: 10.1016/j.ygyno.2011.10.007. Epub 2011 Oct 27. PMID 22035806

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin & Paclitaxel & Radiation: Pelvic Radiation Therapy: Drug:Carboplatin and Paclitaxel and Radiation: Pelvic Radiation Therapy
  Carboplatin and Paclitaxel and Pelvic Radiation Therapy : Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
  Carboplatin and Paclitaxel and Radiation Therapy : Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
Period: Overall Study
Arm/Group | Carboplatin & Paclitaxel & Radiation: Pelvic Radiation Therapy
Started | 81
Completed | 65
Not Completed | 16

BASELINE CHARACTERISTICS:
Population: We considered 72 patients as baseline participants because they are the ones who completed the first three cycles of chemotherapy followed by at least partial RT. Of the 72 patients, 65 of them completed all prescribed regimen of treatment. This was the reason for the discrepancy.
Groups:
- Drug:Carboplatin, Paclitaxel & Radiation: Drug:Carboplatin and Paclitaxel and Radiation: Pelvic Radiation Therapy
  Carboplatin and Paclitaxel and Pelvic Radiation Therapy : Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
  Carboplatin and Paclitaxel and Radiation Therapy : Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
Arm/Group | Drug:Carboplatin, Paclitaxel & Radiation
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] | 67 [43 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Toxicity and Tolerability of Pelvic Radiation "Sandwiched" Between Cycles of Paclitaxel/Carboplatin Chemotherapy in Patients With UPSC
Description: Overall survival analysis of early stage (stage 1 & 2) and late stage (stage 3 & 4)UPSC patients who were prescribed radiation "sanwhiched" between three cycles of paclitaxel/platinum chemotherapy before and after RT. Outcome measures were Progression Free Survival (PFS) and Overall Survival (OS).
Time Frame: Up to 7 years
Population: Kaplan-Meier survival analysis of Progression Free Survival (PFS) and Overall Survival (OS).
Measure: Mean (Standard Error); unit: months
Groups:
- Drug:Carboplatin, Paclitaxel & Radiation: Drug:Carboplatin and Paclitaxel and Radiation: Pelvic Radiation Therapy
  Carboplatin and Paclitaxel and Pelvic Radiation Therapy: Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
  Carboplatin and Paclitaxel and Radiation Therapy: Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
Arm/Group | Drug:Carboplatin, Paclitaxel & Radiation
Number analyzed (Participants) | 72
months
  Early stage (PFS): number analyzed (Participants) | 59
  Early stage (PFS) | 65.5 (3.6)
  Late stage (PFS): number analyzed (Participants) | 13
  Late stage (PFS) | 25.8 (3.0)
  Early stage (OS): number analyzed (Participants) | 59
  Early stage (OS) | 76.5 (4.3)
  Late stage (OS): number analyzed (Participants) | 13
  Late stage (OS) | 35.9 (5.3)

ADVERSE EVENTS:
Time Frame: 435 cycles of paclitaxel/carboplatin were administered on protocol from which frequencies and grades of hematologic and non-hematologic toxicities were tabulated for up to 10 years.
Description: There is no difference in the reporting of adverse events. Adverse even data is not available. Only the toxicity data are available.
Groups:
- Carboplatin & Paclitaxel & Radiation: Pelvic Radiation Therapy: Drug:Carboplatin and Paclitaxel and Radiation: Pelvic Radiation Therapy
  Carboplatin and Paclitaxel and Pelvic Radiation Therapy : Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=6.5) Repeat q 21 days x 3 cycles followed by RT followed by Paclitaxel 175 mg/m2/3 hour & Carboplatin (AUC=5.0)Repeat q 21 days x 3 cycles
  Note: The original PI has left the institution, therefore Dr. Kuo inherited the study. Efforts were made to contact the PI/study team members to locate the raw data, but were unsuccessful. No AE data are available at this time.
Arm/Group | Carboplatin & Paclitaxel & Radiation: Pelvic Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 16/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

LIMITATIONS AND CAVEATS:
There are minor differences in the carboplatin doses between the current trial and our pilot study.

This is a single institution trial. A limited number of advanced stage patients was accrued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes